CLINICAL TRIAL: NCT07259655
Title: Management of Post-Induction Hypotension in Emergency Abdominal Surgery: Norepinephrine Versus Ephedrine
Brief Title: Management of Post-Induction Hypotension in Emergency Abdominal Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: the investigators collected the necessary sample size for the internal validity of the study
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, jebri alia, Head of Anesthesiology and Intensive Care Department at Charles Nicolle Hospital in Tunis, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWA 00032748
Record Dates: First submitted 2025-09-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Post-induction Hypotension
Keywords: norepinephrine; ephedrine; post-induction hypotension; general anesthesia; abdominal emergency
MeSH Terms: interventions — Ephedrine; Norepinephrine

STUDY DESIGN:
Intervention Model Description: This randomized double-blind trial compares diluted norepinephrine (10 µg boluses) versus ephedrine (6 mg boluses) for managing anesthesia-induced hypotension during emergency abdominal surgery. Primary objectives: maintain SBP ≥80% of baseline and compare required bolus numbers. Secondary: incidence of tachycardia (HR >100 bpm), bradycardia (HR <60 bpm) or hypertension. Inclusion: adults >18 years with digestive emergencies (appendicitis, obstruction, etc.), ASA I-III stable. Exclusion: arrhythmias, pulmonary hypertension, septic/hemorrhagic shock. 100 patients randomized to two groups (50 each). Medications prepared in identical syringes (A/B) to maintain blinding.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Ephedrine group) (Active Comparator): Participants receive ephedrine 6 mg IV boluses for the management of anesthesia-induced hypotension during emergency abdominal surgery.
  Interventions: Drug: Ephedrine (6 mg boluses)
- Group 2 (Norepinephrine group) (Active Comparator): Participants receive diluted norepinephrine 10 µg IV boluses for the management of anesthesia-induced hypotension during emergency abdominal surgery.
  Interventions: Drug: Norepinephrine (10 µg boluses)

INTERVENTIONS:
Drug: Ephedrine (6 mg boluses) — Ephedrine 6 mg IV boluses administered when systolic or diastolic blood pressure decreases by ≥20% from baseline. Bolus may be repeated after 1 minute if hypotension persists.
  Arms: Group 1 (Ephedrine group)
Drug: Norepinephrine (10 µg boluses) — Diluted norepinephrine 10 µg IV boluses administered when systolic or diastolic blood pressure decreases by ≥20% from baseline. Bolus may be repeated after 1 minute if hypotension persists.
  Arms: Group 2 (Norepinephrine group)

SUMMARY:
The goal of this clinical trial is to compare the efficacy of two vasopressors (norepinephrine vs. ephedrine) in treating hypotension in adult patients (aged 18+, ASA I-III) undergoing general anesthesia for abdominal surgical emergencies (e.g., appendicitis, intestinal obstruction, peritonitis). The main questions it aims to answer are:

* Which drug is more effective at maintaining intraoperative blood pressure (SBP ≥ 80% of baseline)?
* How many boluses of each vasopressor are required to maintain target blood pressure?

Researchers will compare the norepinephrine group (receiving 10 µg boluses) to the ephedrine group (receiving 6 mg boluses) to see if norepinephrine is superior for maintaining hemodynamic stability and reduces the number of interventions needed.

Participants will:

* Be randomly assigned to receive one of the two study drugs.
* Undergo standard general anesthesia with close hemodynamic monitoring.
* Receive boluses of the assigned vasopressor whenever their blood pressure drops below a predefined threshold.

DETAILED DESCRIPTION:
Post-induction hypotension is a frequent and clinically significant event in patients undergoing emergency abdominal surgery, where baseline hemodynamic instability and reduced physiological reserve are common. The combination of absolute or relative hypovolemia, systemic inflammation, sepsis, and the cardiovascular depressive effects of anesthetic drugs increases the likelihood of early intraoperative hypotension. Preventing and promptly correcting this hemodynamic deterioration is essential, as sustained hypotension has been associated with renal injury, myocardial ischemia, and increased postoperative morbidity.

Ephedrine has historically been used as the first-line agent for anesthesia-induced hypotension because of its mixed α- and β-adrenergic activity. However, concerns regarding tachycardia, variable efficacy, and diminished responsiveness in catecholamine-depleted states have encouraged interest in using diluted norepinephrine as an alternative. Low-dose norepinephrine boluses provide predominantly α-adrenergic vasoconstriction with minimal chronotropic effect, offering a potentially more stable hemodynamic profile. Recent evidence from obstetric and non-obstetric anesthesia suggests that norepinephrine may be effective in restoring blood pressure while reducing heart rate fluctuations.

This randomized double-blind study was designed to compare norepinephrine boluses with ephedrine boluses for the management of anesthesia-induced hypotension in the specific setting of emergency abdominal surgery. The study aims to better characterize the hemodynamic response to each drug in a high-risk population frequently presenting with metabolic disturbances, fluid deficits, and variable sympathetic tone. By evaluating the need for repeated vasopressor administration and the rapidity of blood pressure restoration, the study seeks to determine whether norepinephrine may offer superior intraoperative stability compared with the traditional use of ephedrine. The findings may contribute to optimizing vasopressor strategies in emergency surgical anesthesia and reducing short-term hemodynamic complications.

Conditions Conditions: Post-induction Hypotension Keywords: norepinephrine ephedrine post-induction hypotension general anesthesia abdominal emergency Study Design Study Type: Interventional The intraoperative protocol begins with standard patient preparation including verification of the pre-anesthesia checklist and initiation of monitoring with ECG, pulse oximetry and non-invasive blood pressure measurements at 3minute intervals. Three baseline hemodynamic measurements are recorded and averaged to establish reference values, while two 18G peripheral venous lines are secured for fluid and medication administration. Preload status is assessed using ultrasound measurement of inferior vena cava collapsibility, with crystalloid fluid administration of 10-20 mL/kg initiated if the collapsibility index exceeds 40-50%. Following preoxygenation with 100% FiO2, rapid sequence induction is performed using propofol 2-5 mg/kg and succinylcholine 1 mg/kg, followed by endotracheal intubation confirmed by capnography. Anesthesia maintenance consists of propofol infusion at 6-12 mg/kg/h, fentanyl 2-3 μg/kg for analgesia, and intermittent cisatracurium for neuromuscular blockade, with mechanical ventilation parameters set to 6-8 mL/kg tidal volume and 16-25 breaths per minute targeting end-tidal CO2 of 35-45 mmHg. Hypotension, defined as SBP <90 mmHg, MAP <65 mmHg or a 20% decrease from baseline, is managed with 2 mL boluses of the study drug (either 6 mg ephedrine or 10 μg norepinephrine) repeated after 1 minute if needed, with escalation to norepinephrine infusion at 0.25 mg/mL for refractory cases. Hemodynamic parameters are recorded every 3 minutes for the first 20 minutes post-induction and every 5 minutes thereafter, with documentation of hypotensive episodes, vasopressor requirements, and any adverse hemodynamic events including hypertension, bradycardia or tachycardia. The procedure concludes with extubation when standard criteria are met and transfer to the post-anesthesia care unit for continued monitoring.

Statistical Analysis: Data entry and analysis will be performed using SPSS software (version 25.0). Graphical representations will be prepared using Microsoft Excel 2019.

Descriptive Analysis: Normally distributed continuous quantitative variables will be summarized as mean ± standard deviation. Non-normally distributed continuous variables will be reported as median and interquartile range [IQR: 25%-75%]. Categorical variables will be presented as absolute frequencies (n) and relative frequencies (%).

Analytical Analysis: Associations between two categorical variables will be assessed using Pearson's chi-square test when conditions are met; otherwise, Fisher's exact test will be applied. For comparisons between a categorical and a normally distributed quantitative variable, Student's t-test will be used, while the Mann-Whitney U test will be employed for non-parametric data. A significance level of p < 0.05 will be considered statistically significant. In multivariate analysis, risk estimates will be expressed as odds ratios (OR) with 95% confidence intervals (95% CI).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Digestive emergencies: Appendicitis, cholecystitis, peritonitis, penetrating wounds, strangulated hernia or eventration, intestinal obstruction, complicated diverticulitis, mesenteric ischemia, gastrointestinal perforation.
* Patients classified according to the American Society of Anesthesiologists (ASA) classification as I, II, and stable III

Exclusion Criteria:

* Non-consenting patients.
* Presence of a rhythm disorder.
* Patients with pulmonary hypertension .
* heart failure.
* intra-abdominal hypertension.
* Presence of active bleeding.
* patients using vasopressors at the start of the procedure.
* pregnant women.
* Septic or hemorrhagic shock requiring catecholamines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Rate of restoration of target blood pressure (Efficacy) | Within 3 to 6 minutes post-hypotensive episode
  Percentage of hypotensive episodes where the systolic blood pressure (SBP) was successfully restored to ≥ 80% of the baseline value within the defined time frame.

SECONDARY OUTCOMES:
Number of vasopressor boluses required | Within 3 to 6 minutes post-hypotensive episode
  The total count of vasopressor boluses (norepinephrine or ephedrine) administered to maintain a systolic blood pressure greater than 80% of its baseline value.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Charles Nicolle, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fathy MM, Wahdan RA, Salah AAA, Elnakera AM. Inferior vena cava collapsibility index as a predictor of hypotension after induction of general anesthesia in hypertensive patients. BMC Anesthesiol. 2023 Dec 19;23(1):420. doi: 10.1186/s12871-023-02355-y. PMID 38114949
- [Background] Hassani V, Movaseghi G, Safaeeyan R, Masghati S, Ghorbani Yekta B, Farahmand Rad R. Comparison of Ephedrine vs. Norepinephrine in Treating Anesthesia-Induced Hypotension in Hypertensive Patients: Randomized Double-Blinded Study. Anesth Pain Med. 2018 Aug 26;8(4):e79626. doi: 10.5812/aapm.79626. eCollection 2018 Aug. PMID 30271750
- [Background] Ali Elnabtity AM, Selim MF. Norepinephrine versus Ephedrine to Maintain Arterial Blood Pressure during Spinal Anesthesia for Cesarean Delivery: A Prospective Double-blinded Trial. Anesth Essays Res. 2018 Jan-Mar;12(1):92-97. doi: 10.4103/aer.AER_204_17. PMID 29628561
- [Background] Ngan Kee WD, Lee SWY, Ng FF, Khaw KS. Prophylactic Norepinephrine Infusion for Preventing Hypotension During Spinal Anesthesia for Cesarean Delivery. Anesth Analg. 2018 Jun;126(6):1989-1994. doi: 10.1213/ANE.0000000000002243. PMID 28678073
- [Background] Wong GTC, Irwin MG. Post-induction hypotension: a fluid relationship? Anaesthesia. 2021 Jan;76(1):15-18. doi: 10.1111/anae.15065. Epub 2020 Jul 1. No abstract available. PMID 32609373
- [Background] Bijker JB, van Klei WA, Kappen TH, van Wolfswinkel L, Moons KG, Kalkman CJ. Incidence of intraoperative hypotension as a function of the chosen definition: literature definitions applied to a retrospective cohort using automated data collection. Anesthesiology. 2007 Aug;107(2):213-20. doi: 10.1097/01.anes.0000270724.40897.8e. PMID 17667564